CLINICAL TRIAL: NCT05733208
Title: The Effect of Remote Ischemic Preconditioning on Myocardial Injury After Noncardiac Surgery in Patients at a High Risk of Cardiac Events
Brief Title: The Effect of Remote Ischemic Preconditioning on Myocardial Injury After Noncardiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Zhao, Principal investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E2022236
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Injury; Non-cardiac Surgery; Remote Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Transient ischemic ischemia consisting of 5-minute ischemia followed by 5-minute perfusion will occur on the upper arm
  Interventions: Procedure: Remote ischemic preconditioning
- Sham-remote ischemic preconditioning (Sham Comparator): Transient ischemic ischemia will not actually occur on the upper arm
  Interventions: Procedure: Sham-remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning will consist of four cycles of 5-minute inflation of an blood pressure cuff on the upper arm to 200 mmHg followed by 5-minute deflation. RIPC will be performed twice, one at approximately 24 hours before anaesthesia and the other at approximately 1 hour before anaesthesia.
  Arms: Remote ischemic preconditioning
Procedure: Sham-remote ischemic preconditioning — The identical looking cuff will be placed around the upper arm but not actually inflated for 40 minutes. The control device's components and external appearance are identical to that of the RIPC. However, as compared to the RIPC, the blood pressure cuff's line of inflation is disconnected such that the cuff cannot be inflated. Control treatment will be performed twice, one at approximately 24 hours before anaesthesia and the other at approximately 1 hour before anaesthesia.
  Arms: Sham-remote ischemic preconditioning

SUMMARY:
This is a multicentre, parallel-group, randomised, sham-controlled, observer blinded trial, assessing the efficacy of remote ischemic preconditioning on preventing myocardial injury after noncardiac surgery.

DETAILED DESCRIPTION:
This is a multicentre, randomised, sham-controlled, observer blinded trial. Patients at high clinical risk for cardiovascular events and scheduled to undergo major abdominal surgery will be enrolled. A total of 766 patients are randomised (1:1 ratio) to receive RIPC or no RIPC (control) before anaesthesia induction. RIPC will comprise four alternating cycles of cuff inflation for 5 min to 200 mm Hg and deflation for 5 min. In controls, the identical looking cuff will be placed around the arm but not actually inflated for 40 minutes. The primary outcome was myocardial injury after surgery within three days of surgery. The secondary outcomes were peak plasma hs-cTnT and total hs-cTnT release during the first three days after surgery, hs-cTnT above the prognostically important thresholds, length of hospital stay after surgery, and length of stay in the intensive care unit, myocardial infarction, major adverse cardiovascular events, cardiac-related death and all cause death within 30 days, 6 months, 1 year and 2 years after surgery, postoperative morbidity and adverse events within 30 days after surgery. Besides, blood samples were stored for the other ancillary studies.

ELIGIBILITY:
Inclusion criteria

1. Patients at high clinical risk for cardiovascular events;
2. Patients scheduled to undergo major abdominal surgery.

Exclusion criteria

1. Immediate or urgent surgery or surgery where there is insufficient time to perform RIPC.
2. Abdominal vascular surgery, such as surgery for abdominal aortic aneurysm
3. Experience of conditions precluding the use of RIPC in both arms
4. Patients who are being treated with drugs, such as sulphonamide or nicorandil
5. With contraindications for anaesthetic regimes required in this trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | Within the first three days after surgery
  Number of participants with MINS, diagnosed according to the criteria established by the American Heart Association in 2021

SECONDARY OUTCOMES:
Participants with the concentration of hs-cTnT reaching/above the prognostically important thresholds | Within the first three days after surgery
  Number of participants with the concentration of hs-cTnT reaching/above the prognostically important thresholds
Peak concentration of hs-cTnT within the initial 3 days after surgery | Within the first three days after surgery
  Peak concentration of high-sensitivity cTnT
Total hs-cTnT release within the initial 3 days after surgery (area under the curve) | Within the first three days after surgery
  Total hs-cTnT release
Length of stay in the intensive care unit | expected 2 days after surgery
  Length of intensive care unit stay
Length of postoperative stay | expected 6 days after surgery
  Length of hospital stay after surgery
Myocardial infarction | Within 30 days, 6 months, 1 year and 2 years of surgery
  Number of participants with myocardial infarction
Major adverse cardiovascular events | Within 30 days, 6 months, 1 year and 2 years of surgery
  Cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke
Cardiac-related death | Within 30 days, 6 months, 1 year and 2 years of surgery
  Death related by cardiac reason
All deaths | Within 30 days, 6 months, 1 year and 2 years of surgery
  All-cause death after surgery
Major postoperative morbidity | Within 30 days after surgery
  Major postoperative morbidity
Adverse events | Within 30 days after surgery
  Adverse events

OTHER OUTCOMES:
Acute kidney injury | Within 30 days after surgery
  Acute kidney injury
Postoperative pulmonary complications | Within 30 days after surgery
  Postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Yang Zhao, MD, Principal Investigator — Sixth SunYetSen
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data shown in the tables or figures in the published paper will be shared with other researchers on reasonable requests. Reasonable requests for data sharing should be made to the corresponding author and will be handled in line with the data access and sharing policy of the Human Genetic Resource Administration of China.
Supporting Information: Study Protocol, SAP
Time Frame: from 6 months to 36 months after publication
Access Criteria: Reasonable requests for data sharing should be made to the corresponding author and will be handled in line with the data access and sharing policy of the Human Genetic Resource Administration of China.

REFERENCES:
- [Background] Devereaux PJ, Sessler DI. Cardiac Complications in Patients Undergoing Major Noncardiac Surgery. N Engl J Med. 2015 Dec 3;373(23):2258-69. doi: 10.1056/NEJMra1502824. No abstract available. PMID 26630144
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Smilowitz NR, Berger JS. Perioperative Management to Reduce Cardiovascular Events. Circulation. 2016 Mar 15;133(11):1125-30. doi: 10.1161/CIRCULATIONAHA.115.017787. No abstract available. PMID 26976917
- [Background] Smilowitz NR, Redel-Traub G, Hausvater A, Armanious A, Nicholson J, Puelacher C, Berger JS. Myocardial Injury After Noncardiac Surgery: A Systematic Review and Meta-Analysis. Cardiol Rev. 2019 Nov/Dec;27(6):267-273. doi: 10.1097/CRD.0000000000000254. PMID 30985328
- [Background] Puelacher C, Bollen Pinto B, Mills NL, Duceppe E, Popova E, Duma A, Nagele P, Omland T, Hammerer-Lercher A, Lurati Buse G. Expert consensus on peri-operative myocardial injury screening in noncardiac surgery: A literature review. Eur J Anaesthesiol. 2021 Jun 1;38(6):600-608. doi: 10.1097/EJA.0000000000001486. PMID 33653981
- [Background] Ruetzler K, Smilowitz NR, Berger JS, Devereaux PJ, Maron BA, Newby LK, de Jesus Perez V, Sessler DI, Wijeysundera DN. Diagnosis and Management of Patients With Myocardial Injury After Noncardiac Surgery: A Scientific Statement From the American Heart Association. Circulation. 2021 Nov 9;144(19):e287-e305. doi: 10.1161/CIR.0000000000001024. Epub 2021 Oct 4. PMID 34601955
- [Background] Verbree-Willemsen L, Grobben RB, van Waes JA, Peelen LM, Nathoe HM, van Klei WA, Grobbee DE. Causes and prevention of postoperative myocardial injury. Eur J Prev Cardiol. 2019 Jan;26(1):59-67. doi: 10.1177/2047487318798925. Epub 2018 Sep 12. PMID 30207484
- [Background] Loukogeorgakis SP, Williams R, Panagiotidou AT, Kolvekar SK, Donald A, Cole TJ, Yellon DM, Deanfield JE, MacAllister RJ. Transient limb ischemia induces remote preconditioning and remote postconditioning in humans by a K(ATP)-channel dependent mechanism. Circulation. 2007 Sep 18;116(12):1386-95. doi: 10.1161/CIRCULATIONAHA.106.653782. Epub 2007 Aug 27. PMID 17724264
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384
- [Background] Lau JK, Pennings GJ, Reddel CJ, Campbell H, Liang HPH, Traini M, Gardiner EE, Yong AS, Chen VM, Kritharides L. Remote ischemic preconditioning inhibits platelet alphaIIb beta3 activation in coronary artery disease patients receiving dual antiplatelet therapy: A randomized trial. J Thromb Haemost. 2020 May;18(5):1221-1232. doi: 10.1111/jth.14763. Epub 2020 Mar 13. PMID 32056358
- [Background] Reddel CJ, Pennings GJ, Lau JK, Chen VM, Kritharides L. Circulating platelet-derived extracellular vesicles are decreased after remote ischemic preconditioning in patients with coronary disease: A randomized controlled trial. J Thromb Haemost. 2021 Oct;19(10):2605-2611. doi: 10.1111/jth.15441. Epub 2021 Aug 10. PMID 34196106
- [Background] Crimi G, Pica S, Raineri C, Bramucci E, De Ferrari GM, Klersy C, Ferlini M, Marinoni B, Repetto A, Romeo M, Rosti V, Massa M, Raisaro A, Leonardi S, Rubartelli P, Oltrona Visconti L, Ferrario M. Remote ischemic post-conditioning of the lower limb during primary percutaneous coronary intervention safely reduces enzymatic infarct size in anterior myocardial infarction: a randomized controlled trial. JACC Cardiovasc Interv. 2013 Oct;6(10):1055-63. doi: 10.1016/j.jcin.2013.05.011. PMID 24156966
- [Background] White SK, Frohlich GM, Sado DM, Maestrini V, Fontana M, Treibel TA, Tehrani S, Flett AS, Meier P, Ariti C, Davies JR, Moon JC, Yellon DM, Hausenloy DJ. Remote ischemic conditioning reduces myocardial infarct size and edema in patients with ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt B):178-188. doi: 10.1016/j.jcin.2014.05.015. Epub 2014 Sep 17. PMID 25240548
- [Background] Gaspar A, Lourenco AP, Pereira MA, Azevedo P, Roncon-Albuquerque R Jr, Marques J, Leite-Moreira AF. Randomized controlled trial of remote ischaemic conditioning in ST-elevation myocardial infarction as adjuvant to primary angioplasty (RIC-STEMI). Basic Res Cardiol. 2018 Mar 7;113(3):14. doi: 10.1007/s00395-018-0672-3. PMID 29516192
- [Background] Xie J, Zhang X, Xu J, Zhang Z, Klingensmith NJ, Liu S, Pan C, Yang Y, Qiu H. Effect of Remote Ischemic Preconditioning on Outcomes in Adult Cardiac Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Studies. Anesth Analg. 2018 Jul;127(1):30-38. doi: 10.1213/ANE.0000000000002674. PMID 29210794
- [Background] Jiang Q, Xiang B, Wang H, Huang K, Kong H, Hu S. Remote ischaemic preconditioning ameliorates sinus rhythm restoration rate through Cox maze radiofrequency procedure associated with inflammation reaction reduction. Basic Res Cardiol. 2019 Mar 5;114(3):14. doi: 10.1007/s00395-019-0723-4. PMID 30838448
- [Background] Kosiuk J, Langenhan K, Stegmann C, Uhe T, Dagres N, Dinov B, Kircher S, Richter S, Sommer P, Bertagnolli L, Bollmann A, Hindricks G. Effect of remote ischemic preconditioning on electrophysiological parameters in nonvalvular paroxysmal atrial fibrillation: The RIPPAF Randomized Clinical Trial. Heart Rhythm. 2020 Jan;17(1):3-9. doi: 10.1016/j.hrthm.2019.07.026. Epub 2019 Jul 26. PMID 31356986
- [Derived] Wang F, Liang CJ, Shi JK, Huang QS, Nassirou BM, Wang X, Jin SQ, Zhao Y. Effects of remote ischaemic preconditioning on myocardial injury after major abdominal surgery in patients at high risk for cardiovascular adverse events in China (RIPC-MAS): protocol for a randomised, sham-controlled, observer-blinded trial. BMJ Open. 2023 Jun 23;13(6):e073038. doi: 10.1136/bmjopen-2023-073038. PMID 37355267